CLINICAL TRIAL: NCT04709952
Title: A Clinical Trial Study on the Market to Establish the Safety and Efficacy of a Transcranial DC Stimulation Device in Patients With Depression
Brief Title: Postmarketing Clinical Trial of tDCS to Evaluate Cognitive Ability in Depression Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ji hyun baek, MD, Ph.D (Other)
Responsible Party: Sponsor-Investigator, ji hyun baek, MD, Ph.D, Principal Investigator, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YB_ST_IIT2006
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High real stimulation group (Active Comparator): 2mA tDCS stimulation daily (42 times) for 6 weeks
  Interventions: Device: Transcranial direct current stimulation_High real
- Low real stimulation group (Active Comparator): 1mA tDCS stimulation daily (42 times) for 6 weeks
  Interventions: Device: Transcranial direct current stimulation_Low real
- Sham stimulation group (Sham Comparator): sham stimulation daily (42 times) for 6 weeks
  Interventions: Device: Transcranial direct current stimulation_Sham

INTERVENTIONS:
Device: Transcranial direct current stimulation_High real — Transcranial DCS (tDCS) is applied to patients with depressive disorder taking antidepressants in high real stimulation group (2mA).
  Arms: High real stimulation group
Device: Transcranial direct current stimulation_Low real — Transcranial DCS (tDCS) is applied to patients with depressive disorder taking antidepressants in Low real stimulation group (1mA).
  Arms: Low real stimulation group
Device: Transcranial direct current stimulation_Sham — Transcranial DCS (tDCS) is applied to patients with depressive disorder taking antidepressants in sham stimulation group (0mA).
  Arms: Sham stimulation group

SUMMARY:
This study is a multicenter, double-blind, randomized, and confirmed clinical trial in patients taking antidepressants during the 6-week stimulation period , sham stimulation group, low real stimulation group (1mA), high real stimulation group (2mA) and treatment every day for 6 weeks (a total of 42 times). As a primary outcome, the investigator analyze the improvement effect of working memory ability, and confirm whether the effects of anxiety and depression are improved by the secondary outcome, together with the quality of life evaluation.

DETAILED DESCRIPTION:
During the clinical trial period, a total of 4 to 5 outpatient visits are made, and changes are evaluated through neuropsychological examination by visiting at 2, 4 and 6 weeks based on the baseline time point. In addition, in the case of patients who agree after 6 weeks of participation, an additional 6 weeks of high real stimulation is used to conduct an open extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of major depressive disorder
2. CGI severity (severity of Illness) score of 3 or higher
3. Patients receiving medication for depression at the time of study participation
4. Those who can read and understand the subject's explanation and consent form and who can respond to questionnaires

Exclusion Criteria:

1. History of clinically significant medical neurological disease or history of head injury
2. In case of mental retardation or cognitive impairment enough to affect the writing of consent form or conducting research
3. Severe suicidal risk or psychotic symptoms determined by the clinician
4. In the case of a contraindication to the implementation of tDCS (when a metallic auxiliary tool is inserted in the head)
5. Those who are judged to have problems with the attachment of EEG and DC stimulation electrodes due to deformities, inflammatory reactions, or other dermatological problems at the electrode attachment site
6. Among female subjects who are likely to become pregnant, those who do not agree to contraception by a medically acceptable method for up to 24 weeks after application of the investigational medical device in this clinical trial
7. Pregnant women
8. Any other person who has reasons to judge that the investigator is unsuitable for participation in the clinical trial

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Working memory ability evaluation(N-Back tast) | Change from Baseline Working memory ability evaluation at 6 weeks.
  N-back tasks are continuous-recognition measures that present stimulus sequences, such as letters or pictures; for each item in the sequence, people judge whether it matches the one presented n items ago. As the number of correct answers increases, it means improvement in cognitive function.

SECONDARY OUTCOMES:
Hamilton Rating Scale | Change from Baseline Hamilton Rating Scale evaluation at 2,4,6 weeks
  The patient is rated by a clinician on 17 items scored either on a 3-point or 5-point Likert-type scale. The lower the total score, the better the symptoms.
Hamilton Anxiety Rating Scale | Change from Baseline Hamilton Anxiety Rating Scale evaluation at 2,4,6 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. Upon the completion of the evaluation, the clinician compiles a total, composite score based upon the summation of each of the 14 individually rated items. This calculation will yield a comprehensive score in the range of 0 to 56. It has been predetermined that the results of the evaluation can be interpreted as follows. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity.The lower the total score, the better the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hyun Baek, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Lee CW, Park K, Ahn JE, Jang Y, Park YS, Yu H, Lee D, Ihm HK, Lee J, Kim J, Lee YI, Lim SE, Kwon SS, Park HY, Ha TH, Yoon IY, Myung W, Baek JH. Efficacy and safety of home-based transcranial direct current stimulation as adjunct treatment for cognitive improvement in major depressive disorder: A double-blind, randomized, multi-site clinical trial. Eur Psychiatry. 2025 Jan 15;68(1):e15. doi: 10.1192/j.eurpsy.2024.1811. PMID 39809704